CLINICAL TRIAL: NCT06901830
Title: A PhaseⅡ, Randomized, Double-Blind, Placebo- and Active- Controlled Study of YZJ-4729 Tartrate Injection for the Treatment of Moderate to Severe Pain After Orthopedic Surgery
Brief Title: A Study of YZJ-4729 Tartrate Injection for the Treatment of Pain After Orthopedic Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YZJ-4729-2-02
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental Group 1 (Experimental)
  Interventions: Drug: YZJ-4729
- Experimental Group 2 (Experimental)
  Interventions: Drug: YZJ-4729
- Experimental Group 3 (Experimental)
  Interventions: Drug: YZJ-4729
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo Comparator: Saline
- Active Comparator (Active Comparator)
  Interventions: Drug: Active Comparator: Morphine

INTERVENTIONS:
Drug: YZJ-4729 — Loading dose + demand dose
  Arms: Experimental Group 1; Experimental Group 2; Experimental Group 3
Drug: Placebo Comparator: Saline — Loading dose + demand dose
  Arms: Placebo Comparator
Drug: Active Comparator: Morphine — Loading dose + demand dose
  Arms: Active Comparator

SUMMARY:
The primary objective is to evaluate the analgesic efficacy and safety of IV YZJ-4729 Tartrate Injection in patients with acute postoperative pain following Orthopedic surgery

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand the study purpose and cooperate with the study procedures of this trial, voluntarily provide written informed consent
2. BMI≥18.0 kg/m2 and ≤28.0 kg/m2
3. ASA I to II
4. Experiences a pain intensity rating of moderate to severe acute pain following orthopedic surgery, with a pain intensity score of ≥4 on a Numeric Rating Scale (NRS) within 4 hours post-surgery

Exclusion Criteria:

1. Opioid allergy
2. Nervous system diseases (e.g. epilepsy)
3. Psychiatric disorders (e.g. depression)
4. History of difficult airways
5. Random blood glucose ≥11.1 mmol/L
6. Subjects with systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg or systolic blood pressure < 90 mmHg
7. Abnormal pulse oxygen saturation (SpO2 <92 %)
8. Abnormal liver function or renal function
9. Used agents that could affect the analgesic response
10. Used agents that could affect drug metabolism
11. Has previously participated in another YZJ-4729 clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The sum of pain intensity differences in pain score over 48 hours at rest | 48 hours
  Pain intensity will be evaluated using an 11-point (0-10) Numeric Pain Rating Scale (NRS), with higher numbers indicating a higher pain intensity, administered over 48 hours.

SECONDARY OUTCOMES:
The time of first using of rescue analgesics | 0-48 hours
The proportion of subjects using rescue analgesics | 0-48 hours
The number of times for rescue analgesics using | 0-48 hours
The cumulative dose used of rescue analgesics | 0-48 hours
The resting Sum of Pain Intensity Differences Over 12,24,24~48 | 0-48 hours
The active Sum of Pain Intensity Differences Over 12,24,48,24~48 | 0-48 hours
Participant satisfaction scores for analgesia treatment | 48 hours
  Participants recalled the postoperative analgesia effect and rated their satisfaction on a scale of 1 to 5, with 1 representing dissatisfied and 5 representing very satisfied
Investigator satisfaction scores for analgesia treatment | 48 hours
  Postoperative analgesia was evaluated by investigators. The scale ranges from 1 to 5, with 1 being dissatisfied and 5 being very satisfied

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - The Third Xiangya Hospital of Central South University, Changsha
  - Chengdu Second People's Hospital, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - The Third People's Hospital of Chengdu, Chengdu
  - The First Hospital of Jilin University, Ch’ang-ch’un
  - Dalian University Affiliated Zhongshan Hospital, Dalian
  - Dongguan People's Hospital, Dongguan
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - The Second People's Hospital of Hefei, Hefei
  - Jinhua Central Hospital, Jinhua
  - Mianyang Central Hospital, Mianyang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - The Third Hospital of Hebei Medical University, Shijiazhuang
  - Suzhou University Affiliated Second Hospital, Suzhou
  - Henan Provincial People's Hospital, Zhengzhou